CLINICAL TRIAL: NCT03701334
Title: A Phase III Multi-center, Randomized, Open-label Trial to Evaluate Efficacy and Safety of Ribociclib With Endocrine Therapy as an Adjuvant Treatment in Patients With Hormone Receptor-positive, HER2-negative Early Breast Cancer (New Adjuvant TriAl With Ribociclib [LEE011]: NATALEE)
Brief Title: A Trial to Evaluate Efficacy and Safety of Ribociclib With Endocrine Therapy as Adjuvant Treatment in Patients With HR+/HER2- Early Breast Cancer
Acronym: NATALEE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Translational Research in Oncology (Other)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLEE011O12301C; 2023-510357-42-00 (Registry Identifier: EU CT Number)
Expanded Access: NCT05038631 (Available)
Record Dates: First submitted 2018-09-21; First posted 2018-10-10 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Early Breast Cancer
Keywords: early breast cancer (EBC); HR+/HER2-; adjuvant; LEE011; ribociclib; CDK4/6 inhibitor
MeSH Terms: conditions — Breast Neoplasms | interventions — ribociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ribociclib + Endocrine Therapy (Experimental): Participants will receive ribociclib 400 mg once daily on days 1-21 of a 28-day cycle and endocrine therapy once daily continuously
  Interventions: Drug: Ribociclib; Other: Endocrine Therapy
- Endocrine Therapy (Active Comparator): Participants will receive endocrine therapy only once daily continuously
  Interventions: Other: Endocrine Therapy

INTERVENTIONS:
Drug: Ribociclib — Ribociclib orally taken at 400 mg on days 1 to 21 of a 28-day cycle
  Arms: Ribociclib + Endocrine Therapy
Other: Endocrine Therapy — ET will be administered according to the local clinical guidelines and current local prescribing information

SUMMARY:
A phase III multi-center, randomized, open-label trial to evaluate efficacy and safety of ribociclib with endocrine therapy as adjuvant treatment in patients with HR+/HER2- Early Breast Cancer (EBC)

DETAILED DESCRIPTION:
The trial will include pre and postmenopausal women and men with HR-positive, HER2-negative EBC, with an Anatomic Stage Group III, IIB or a subset of Stage IIA cases, after adequate surgical resection, radiotherapy (if indicated), adjuvant or neoadjuvant chemotherapy (if indicated), and who are deemed to be eligible for adjuvant ET for at least 60 months of duration.

Approximately 5,000 patients will be randomized (using an Interactive Response Technology system [IRT]) into two treatment arms in a 1:1 ratio.

The trial will include screening, treatment, and follow up phases.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 18 years-old at the time of PICF signature
* Patient is female with known menopausal status at the time of randomization or initiation of adjuvant ET (whichever occurs earlier), or male.
* Patient with histologically confirmed unilateral primary invasive adenocarcinoma of the breast with a date of initial cytologic or histologic diagnosis within 18 months prior to randomization.
* Patient has breast cancer that is positive for ER and/or PgR
* Patient has HER2-negative breast cancer
* Patient has available archival tumor tissue from the surgical specimen
* Patient after surgical resection where tumor was removed completely, with the final surgical specimen microscopic margins free from tumor, and belongs to one of the following categories: anatomic stage group II or III
* If indicated, patient has completed adjuvant and/or neoadjuvant chemotherapy according to the institutional guidelines
* If indicated, patient has completed adjuvant radiotherapy according to the institutional guidelines
* Patient has an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Patient has no contraindication for the adjuvant ET in the trial and is planned to be treated with ET for 5 years

Exclusion Criteria:

* Patient has received any CDK4/6 inhibitor
* Patient has received prior treatment with tamoxifen, raloxifene or AIs for reduction in risk ("chemoprevention") of breast cancer and/or treatment for osteoporosis within the last 2 years prior to randomization. Patient is concurrently using hormone replacement therapy.
* Patient has received prior treatment with anthracyclines at cumulative doses of 450 mg/m² or more for doxorubicin, or 900 mg/m² or more for epirubicin.
* Patient with a known hypersensitivity to any of the excipients of ribociclib and/or ET
* Patient with distant metastases of breast cancer beyond regional lymph nodes (stage IV according to AJCC 8th edition) and/or evidence of recurrence after curative surgery.
* Patient is concurrently using other anti-neoplastic therapy with the exception of adjuvant ET
* Patient has had major surgery, chemotherapy or radiotherapy within 14 days prior to randomization
* Patient has not recovered from clinical and laboratory acute toxicities related to prior anti-cancer therapies
* Patient has a concurrent invasive malignancy or a prior invasive malignancy whose treatment was completed within 2 years before randomization
* Patient has known HIV infection, Hepatitis B or C infection
* Clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormality
* Patient is currently receiving any of the following substances within 7 days before randomization - Concomitant medications, herbal supplements, and/or fruits that are known as strong inhibitors or inducers of CYP3A4/5 or Medications that have a narrow therapeutic window and are predominantly metabolized through CYP3A4/5
* is currently receiving or has received systemic corticosteroids ≤ 2 weeks prior to starting trial treatment
* Patient has impairment of GI function or GI disease that may significantly alter the absorption of the oral trial treatments
* Patient has any other concurrent severe and/or uncontrolled medical condition that would, in the Investigator's judgment, cause unacceptable safety risks, contraindicate patient participation in the clinical trial or compromise compliance with the protocol
* Participation in other studies involving investigational drug(s) within 30 days prior to randomization or within 5 half-lives of the investigational drug(s) (whichever is longer), or participation in any other type of medical research judged not to be scientifically or medically compatible with this trial.
* Pregnant or breast-feeding (lactating) women or women who plan to become pregnant or breast-feed during the trial

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5101 (Actual)
Dates: Start 2018-12-07 (Actual); Primary Completion 2026-05-29 (Estimated); Study Completion 2026-05-29 (Estimated)

PRIMARY OUTCOMES:
Invasive Disease-Free Survival (iDFS) | Up to approximately 91 months
  iDFS using STEEP criteria (Standardized Definitions for Efficacy End Points in Adjuvant Breast Cancer Trials), as assessed by Investigator. iDFS is defined as time from the date of randomization to the date of the first event of local invasive breast recurrence, regional invasive recurrence, distant recurrence, death (any cause), contralateral invasive BC, or second primary non-breast invasive cancer (excluding basal and squamous cell carcinomas of the skin).

SECONDARY OUTCOMES:
Recurrence-free survival (RFS) | Up to approximately 91 months
  RFS using STEEP criteria (Standardized Definitions for Efficacy End Points in Adjuvant Breast Cancer Trials). RFS is defined as the time from date of randomization to date of first event of local invasive breast recurrence, regional invasive recurrence, distant recurrence, or death (any cause).
Distant disease-free survival (DDFS) | Up to approximately 91 months
  DDFS using STEEP criteria. DDFS is defined as the time from date of randomization to date of first event of distant recurrence, death (any cause), or second primary non-breast invasive cancer (excluding basal and squamous cell carcinomas of the skin).
Overall Survival (OS) | Up to approximately 91 months
  OS is defined as the time from date of randomization to date of death due to any cause.
Change from baseline in the global health status Quality of life scale score as assessed by EORTC QLQ-C30 | Up to approximately 91 months
  The EORTC QLQ-C30 contains functional scales, symptom scales, single items scale and a global health status/QoL scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Change from baseline in the physical functioning sub-scale score as assessed by EORTC QLQ-C30 | Up to approximately 91 months
  The EORTC QLQ-C30 contains functional scales, symptom scales, single items scale and a global health status/QoL scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
PK parameters: Ctrough and other applicable parameters for ribociclib | Cycle 1 Day 15
  Pharmacokinetics of ribociclib: Ctrough and other applicable parameters

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (344):
- United States (73):
  - University of Alabama at Birmingham-Kirklin Clinic, Birmingham, Alabama
  - Cancer Treatment Centers of America, Goodyear, Arizona
  - St Bernards Medical Center, Jonesboro, Arkansas
  - Comprehensive Blood and Cancer, Bakersfield, California
  - UCLA Beverly Hills, Beverly Hills, California
  - UCLA Burbank, Burbank, California
  - Encino Research Center, Encino, California
  - St. Jude Heritage Medical Group, Fullerton, California
  - UCLA Hematology Oncology, Laguna Hills, California
  - Southern CA Oncology Rsrch Alliance, Los Angeles, California
  - Stanford University Medical Center, Palo Alto, California
  - UCLA Pasadena HC Hemato Onco, Pasadena, California
  - UCLA Porter Ranch Hemato and Onco, Porter Ranch, California
  - Cancer Care Associates Medical Grp, Redondo Beach, California
  - Sharp Memorial Hospital, San Diego, California
  - UCSF, San Francisco, California
  - Central Coast Medical Oncology Corporation, Santa Maria, California
  - UCLA Santa Monica Hematology Oncology, Santa Monica, California
  - Lundquist Inst BioMed at Harbor, Torrance, California
  - UCLA Valencia, Valencia, California
  - Valley Breast Care, Van Nuys, California
  - UCLA Cancer Center Westlake Village, Westlake Village, California
  - University Of Colorado Hospital, Aurora, Colorado
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Hospital of Central Connecticut, New Britain, Connecticut
  - Yale University School Of Medicine, New Haven, Connecticut
  - Norwalk Hospital, Norwalk, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Holy Cross Hospital-Ft. Lauderdale, Fort Lauderdale, Florida
  - Florida Cancer Specialists, Fort Myers, Florida
  - Memorial Cancer Institute, Hollywood, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Orlando Health Clinical Trials, Orlando, Florida
  - Florida Cancer Specialists-North, St. Petersburg, Florida
  - Florida Cancer Specialists Pan, Tallahassee, Florida
  - Florida Cancer Specialists, West Palm Beach, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Southeastern Regional Medical Center, Newnan, Georgia
  - Cancer Treatment Centers of America, Zion, Illinois
  - Cancer Care Center, New Albany, Indiana
  - University of Kansas Cancer Center, Westwood, Kansas
  - Cancer Center of Kansas, Wichita, Kansas
  - Norton Cancer Institute, Louisville, Kentucky
  - Mercy Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan Cancer Center, Ann Arbor, Michigan
  - Fairview Health Services, Maple Grove, Minnesota
  - Metro Minnesota CCOP, Saint Louis Park, Minnesota
  - Park Nicollet Institute, Saint Louis Park, Minnesota
  - Saint Lukes Hospital of Kansas City, Kansas City, Missouri
  - HCA Midwest Division, Kansas City, Missouri
  - David C Pratt Cancer Center, St Louis, Missouri
  - St Vincent Frontier Cancer Center, Billings, Montana
  - Saint Francis Medical Center, Grand Island, Nebraska
  - Comprehensive Cancer Cntr Of Nevada, Henderson, Nevada
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Perlmutter Cancer Centre, New York, New York
  - Randolph Medical Associates, Asheboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Kaiser Permanente NW Region, Clackamas, Oregon
  - Penn State Hershey Cancer Institute, Hershey, Pennsylvania
  - Cancer Treatment Centers of America Eastern Regional Medical Center, Philadelphia, Pennsylvania
  - The West Clinic, Germantown, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Baylor Charles A Sammons Cancer Cnt, Dallas, Texas
  - Ctr For Cancer And Blood Disorders, Fort Worth, Texas
  - MD Anderson Cancer Center University of Texas, Houston, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - University of Wisconsin Paul P Carbone Comp Cancer Center, Madison, Wisconsin
- Argentina (8):
  - Novartis Investigative Site, San Salvador de Jujuy, Jujuy Province
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, Rosario, Sante Fe
  - Novartis Investigative Site, San Miguel Tucuman, Tucumán Province
  - Novartis Investigative Site, Rio Negro, Viedma
  - Novartis Investigative Site, CABA
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, La Rioja
- Australia (24):
  - Novartis Investigative Site, Campbelltown, New South Wales
  - Novartis Investigative Site, Coffs Harbour, New South Wales
  - Novartis Investigative Site, Darlinghurst, New South Wales
  - Novartis Investigative Site, Kingswood, New South Wales
  - Novartis Investigative Site, Kogarah, New South Wales
  - Novartis Investigative Site, North Ryde, New South Wales
  - Novartis Investigative Site, St Leonards, New South Wales
  - Novartis Investigative Site, Wahroonga, New South Wales
  - Novartis Investigative Site, Westmead, New South Wales
  - Novartis Investigative Site, Auchenflower, Queensland
  - Novartis Investigative Site, Birtinya, Queensland
  - Novartis Investigative Site, Wooloongabba, Queensland
  - Novartis Investigative Site, Bedford Park, South Australia
  - Novartis Investigative Site, Bendigo, Victoria
  - Novartis Investigative Site, East Melbourne, Victoria
  - Novartis Investigative Site, Epping, Victoria
  - Novartis Investigative Site, Fitzroy, Victoria
  - Novartis Investigative Site, Franston, Victoria
  - Novartis Investigative Site, Heidelberg, Victoria
  - Novartis Investigative Site, Melbourne, Victoria
  - Novartis Investigative Site, Shepparton, Victoria
  - Novartis Investigative Site, Murdoch, Western Australia
  - Novartis Investigative Site, Nedlands, Western Australia
  - Novartis Investigative Site, Liverpool
- Austria (5):
  - Novartis Investigative Site, Innsbruck, Tyrol
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Vienna
- Belgium (11):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Charleroi
  - Novartis Investigative Site, Edegem
  - Novartis Investigative Site, Hasselt
  - Novartis Investigative Site, Jette
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Libramont
  - Novartis Investigative Site, Liège
  - Novartis Investigative Site, Namur
  - Novartis Investigative Site, Wilrijk
  - Novartis Investigative Site, Yvoir
- Brazil (13):
  - Novartis Investigative Site, Londrina, Paraná
  - Novartis Investigative Site, Ijuí, Rio Grande do Sul
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Barretos, São Paulo
  - Novartis Investigative Site, Santo André, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, Caxias do Sul
  - Novartis Investigative Site, Passo Fundo
  - Novartis Investigative Site, Piracicaba
  - Novartis Investigative Site, Recife
  - Novartis Investigative Site, Rio de Janeiro
  - Novartis Investigative Site, Salvador
  - Novartis Investigative Site, São Paulo
- Canada (20):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Kelowna, British Columbia
  - Novartis Investigative Site, North Vancouver, British Columbia
  - Novartis Investigative Site, Surrey, British Columbia
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, Greater Sudbury, Ontario
  - Novartis Investigative Site, Kitchener, Ontario
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Newmarket, Ontario
  - Novartis Investigative Site, Oshawa, Ontario
  - Novartis Investigative Site, Sault Ste. Marie, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Windsor, Ontario
  - Novartis Investigative Site, Fleurimont, Quebec
  - Novartis Investigative Site, Greenfield Park, Quebec
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
  - Novartis Investigative Site, Saint-Jérôme, Quebec
- China (15):
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Shijiazhuang, Hebei
  - Novartis Investigative Site, Harbin, Heilongjiang
  - Novartis Investigative Site, Zhengzhou, Henan
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Suzhou, Jiangsu
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Chongqing
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Tianjin
  - Novartis Investigative Site, Zhenjiang
- France (27):
  - Novartis Investigative Site, Nice, Alpes Maritimes
  - Novartis Investigative Site, Dijon, Cote D Or
  - Novartis Investigative Site, Limoges, Haute Vienne
  - Novartis Investigative Site, Saint-Cloud, Hauts De Seine
  - Novartis Investigative Site, Rennes, Ille Et Vilaine
  - Novartis Investigative Site, Grenoble, Isere
  - Novartis Investigative Site, Lyon, Rhone
  - Novartis Investigative Site, Amiens
  - Novartis Investigative Site, Angers
  - Novartis Investigative Site, Argenteuil
  - Novartis Investigative Site, Avignon
  - Novartis Investigative Site, Besançon
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Bron
  - Novartis Investigative Site, Caen
  - Novartis Investigative Site, Le Mans
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pierre-Bénite
  - Novartis Investigative Site, Rouen
  - Novartis Investigative Site, Saint-Herblain
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Vandœuvre-lès-Nancy
  - Novartis Investigative Site, Villejuif
- Germany (27):
  - Novartis Investigative Site, Ravensburg, Baden-Wurttemberg
  - Novartis Investigative Site, Munich, Bavaria
  - Novartis Investigative Site, Würzburg, Bavaria
  - Novartis Investigative Site, Cottbus, Brandenburg
  - Novartis Investigative Site, Frankfurt am Main, Hesse
  - Novartis Investigative Site, Georgsmarienhütte, Lower Saxony
  - Novartis Investigative Site, Hanover, Lower Saxony
  - Novartis Investigative Site, Essen, North Rhine-Westphalia
  - Novartis Investigative Site, Mönchengladbach, North Rhine-Westphalia
  - Novartis Investigative Site, Velbert, North Rhine-Westphalia
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Bad Liebenwerda
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Bottrop
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Mannheim
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Regensburg
  - Novartis Investigative Site, Schweinfurt
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Ulm
- Hungary (9):
  - Novartis Investigative Site, Zalaegerszeg, Zala County
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Kecskemét
  - Novartis Investigative Site, Pécs
  - Novartis Investigative Site, Szeged
  - Novartis Investigative Site, Szekszárd
  - Novartis Investigative Site, Szombathely
  - Novartis Investigative Site, Tatabánya
- Ireland (4):
  - Novartis Investigative Site, Wilton, Cork
  - Novartis Investigative Site, County Limerick
  - Novartis Investigative Site, Dublin
  - Novartis Investigative Site, Waterford
- Italy (11):
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Catania, CT
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Palermo, PA
  - Novartis Investigative Site, Aviano, PN
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Candiolo, TO
  - Novartis Investigative Site, Napoli
- Poland (13):
  - Novartis Investigative Site, Warsaw, Ul Roentgena 5
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Gdynia
  - Novartis Investigative Site, Gliwice
  - Novartis Investigative Site, Grudziądz
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Lublin
  - Novartis Investigative Site, Opole
  - Novartis Investigative Site, Ostrołęka
  - Novartis Investigative Site, Otwock
  - Novartis Investigative Site, Wieliszew
  - Novartis Investigative Site, Wroclaw
- Romania (4):
  - Novartis Investigative Site, Craiova, Dolj
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Cluj-Napoca
  - Novartis Investigative Site, Timișoara
- Russia (17):
  - Novartis Investigative Site, Kazan', Russian Federation
  - Novartis Investigative Site, Saint Petersburg, Sankt-Peterburg
  - Novartis Investigative Site, Chelyabinsk
  - Novartis Investigative Site, Kostroma
  - Novartis Investigative Site, Krasnoyarsk
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Nizhny Novgorod
  - Novartis Investigative Site, Novosibirsk
  - Novartis Investigative Site, Obninsk
  - Novartis Investigative Site, Omsk
  - Novartis Investigative Site, Orenburg
  - Novartis Investigative Site, Rostov-on-Don
  - Novartis Investigative Site, Ryazan
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Tyumen
  - Novartis Investigative Site, Ufa
  - Novartis Investigative Site, Yaroslavl
- South Korea (11):
  - Novartis Investigative Site, Seoul, Daegu
  - Novartis Investigative Site, Wŏnju, Gangwon-do
  - Novartis Investigative Site, Bundang Gu, Gyeonggi-do
  - Novartis Investigative Site, Suwon, Gyeonggi-do
  - Novartis Investigative Site, Gyeonggi-do, Korea
  - Novartis Investigative Site, Cheongju-si, North Chungcheong
  - Novartis Investigative Site, Seoul, Seocho Gu
  - Novartis Investigative Site, Incheon
  - Novartis Investigative Site, Seongnam
  - Novartis Investigative Site, Seoul
  - Novartis Investigative Site, Ulsan
- Spain (39):
  - Novartis Investigative Site, Elche, Alicante
  - Novartis Investigative Site, Granada, Andalusia
  - Novartis Investigative Site, Huelva, Andalusia
  - Novartis Investigative Site, Jaén, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Vitoria-Gasteiz, Araba
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, Manresa, Barcelona
  - Novartis Investigative Site, Sabadell, Barcelona
  - Novartis Investigative Site, Donostia / San Sebastian, Basque Country
  - Novartis Investigative Site, Bilbao, Bizkaia
  - Novartis Investigative Site, Salamanca, Castille and León
  - Novartis Investigative Site, Badalona, Catalonia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Badajoz, Extremadura
  - Novartis Investigative Site, Cáceres, Extremadura
  - Novartis Investigative Site, Lugo, Galicia
  - Novartis Investigative Site, Fuenlabrada, Madrid
  - Novartis Investigative Site, Majadahonda, Madrid
  - Novartis Investigative Site, El Palmar, Murcia
  - Novartis Investigative Site, Pamplona, Navarre
  - Novartis Investigative Site, Vigo, Pontevedra
  - Novartis Investigative Site, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Novartis Investigative Site, Alicante, Valencia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, A Coruña
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Burgos
  - Novartis Investigative Site, Castellon
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, Girona
  - Novartis Investigative Site, Granada
  - Novartis Investigative Site, Las Palmas GC
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Málaga
  - Novartis Investigative Site, Murcia
  - Novartis Investigative Site, Seville
  - Novartis Investigative Site, Valencia
  - Novartis Investigative Site, Zaragoza
- Taiwan (5):
  - Novartis Investigative Site, Changhua
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Tainan
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District
- United Kingdom (8):
  - Novartis Investigative Site, Truro, Cornwall
  - Novartis Investigative Site, Sutton, Surrey
  - Novartis Investigative Site, Cardiff
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Nottingham
  - Novartis Investigative Site, Oxford
  - Novartis Investigative Site, Preston
  - Novartis Investigative Site, Stoke-on-Trent

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Fasching PA, Stroyakovskiy D, Yardley DA, Huang CS, Crown J, Bardia A, Chia S, Im SA, Martin M, Xu B, Loi S, Barrios C, Untch M, Moroose R, Visco F, Hortobagyi GN, Slamon DJ, Fresco R, Zarate JP, Li Z, Waters S, Hurvitz SA. Ribociclib Plus Endocrine Therapy in Hormone Receptor-Positive/ERBB2-Negative Early Breast Cancer: 4-Year Outcomes From the NATALEE Randomized Clinical Trial. JAMA Oncol. 2025 Nov 1;11(11):1364-1372. doi: 10.1001/jamaoncol.2025.3700. PMID 40996773
- [Derived] Slamon D, Lipatov O, Nowecki Z, McAndrew N, Kukielka-Budny B, Stroyakovskiy D, Yardley DA, Huang CS, Fasching PA, Crown J, Bardia A, Chia S, Im SA, Ruiz-Borrego M, Loi S, Xu B, Hurvitz S, Barrios C, Untch M, Moroose R, Visco F, Afenjar K, Fresco R, Severin I, Ji Y, Ghaznawi F, Li Z, Zarate JP, Chakravartty A, Taran T, Hortobagyi G. Ribociclib plus Endocrine Therapy in Early Breast Cancer. N Engl J Med. 2024 Mar 21;390(12):1080-1091. doi: 10.1056/NEJMoa2305488. PMID 38507751
- [Derived] Slamon DJ, Fasching PA, Hurvitz S, Chia S, Crown J, Martin M, Barrios CH, Bardia A, Im SA, Yardley DA, Untch M, Huang CS, Stroyakovskiy D, Xu B, Moroose RL, Loi S, Visco F, Bee-Munteanu V, Afenjar K, Fresco R, Taran T, Chakravartty A, Zarate JP, Lteif A, Hortobagyi GN. Rationale and trial design of NATALEE: a Phase III trial of adjuvant ribociclib + endocrine therapy versus endocrine therapy alone in patients with HR+/HER2- early breast cancer. Ther Adv Med Oncol. 2023 May 29;15:17588359231178125. doi: 10.1177/17588359231178125. eCollection 2023. PMID 37275963